CLINICAL TRIAL: NCT02920021
Title: Placebo-Controlled Proof of Concept Study to Investigate ANB020 Activity in Adult Patients With Peanut Allergy
Brief Title: Study to Investigate Etokimab (ANB020) Activity in Adult Participants With Peanut Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB020-003
Record Dates: First submitted 2016-09-26; First posted 2016-09-30 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etokimab (Experimental): Participants received a single dose of 300 milligrams (mg) etokimab administered by 1-hour intravenous (IV) infusion on Day 1.
  Interventions: Drug: Etokimab
- Placebo (Placebo Comparator): Participants received a single dose of placebo administered by 1-hour IV infusion on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etokimab — Humanized monoclonal antibody, administered by intravenous infusion
  Other Names: ANB020
  Arms: Etokimab
Drug: Placebo — Administered by intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine etokimab safety, tolerability and activity in adult participants with peanut allergy.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, proof of concept study to assess the safety and tolerability of etokimab in adult participants with peanut allergy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with age > 18 years and able to give informed consent.
* Participants with a confirmed clinically allergic response to peanut.
* Positive clinical reaction during the peanut oral food challenge and no clinical reaction during the placebo challenge
* Positive peanut allergy skin prick test > 3 millimeters (mm) of the negative control and detectable serum peanut-specific Immunoglobulin E (IgE) levels by ImmunoCAP testing.
* Body mass index (BMI) of 18 to 36 kilogram per square meter (kg/m^2) inclusive) and total body weight > 50 kg (110 lb). BMI = weight (kg)/(height [m^2]).
* Willing and able to comply with the study protocol requirements.
* Have the ability to read and understand the study procedures and have the ability to communicate meaningfully with the Investigator and staff.
* Women of childbearing potential, must have a negative serum pregnancy test at screening and Day 1, and be surgically sterile or using an acceptable method of contraception throughout the study and for 15 weeks after the last administration of investigational product. Postmenopausal participants defined as (1) aged over 45 years with at least 1 year of amenorrhea and levels of follicle stimulating hormone over 20 international units per liter (IU/L) or (2) aged over 50 years with at least 1 year of amenorrhea.
* Male participants must be willing to use effective methods of contraception during the entire study period and for 15 weeks after the last administration of investigational product.

Exclusion Criteria:

* Have concomitant dermatological or medical condition(s) which may interfere with the Investigator's ability to evaluate the participant's response to the investigational product.
* Have experienced severe life-threatening anaphylactic reactions to peanuts within 6 months before screening (i.e., requiring an intensive care unit [ICU] admission).
* Positive clinical reaction observed during the placebo oral food challenge.
* Participation in any interventional study for the treatment of peanut and/or food allergies in the 12 months before screening.
* Have received any investigational product or been part of any interventional clinical study within a period of 3 months or 5 half-lives (whichever is longer) before screening.
* Have received systemic corticosteroids, nonsteroidal, immunosuppressant, or immunomodulating drugs treatments within 2 weeks before screening.
* Use of beta blockers, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, or calcium channel blockers within 2 weeks before screening.
* History of ischemic cardiovascular diseases.
* Use of biologics within 6 months before screening or participant is in build-up phase of allergen immunotherapy (excluding peanut) and has not reached maintenance dose.
* Have received antibiotic treatment within 1 week before screening.
* Have a history of hypersensitivity or allergic reactions following infusions of human blood or blood components.
* Have a history of hypersensitivity or allergic reactions a component of etokimab formulation or the inactive ingredients (excipients).
* If female, are pregnant or lactating, or intend to become pregnant during the study period.
* Current diagnosis of asthma requiring Global Initiative for Asthma Assessment (GINA) Step 4 or higher treatment or asthma partially controlled or uncontrolled according to GINA classifications in the last three months before screening.
* History of a life threatening asthma attack within 1 year before screening (example: requiring an intensive care unit admission, intubation with mechanical ventilation).
* Other significant medical conditions that in the opinion of the Principal Investigator, prevent participation in the study.
* History of drug, alcohol or other substance abuse, or other factors limiting the ability to cooperate and to comply with the study protocol.
* Have any other physical, mental, or medical conditions which, in the opinion of the Investigator, make study participation inadvisable or could confound study assessments.
* Receipt of a live attenuated vaccine within 4 weeks before screening.
* Planned surgery during the study or 30 days before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Randazzo, MD, Study Director — AnaptysBio, Inc.
Locations (2):
- United States (2):
  - Stanford Univ. Medical Center, Palo Alto, California
  - Asthma, Inc Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chinthrajah S, Cao S, Liu C, Lyu SC, Sindher SB, Long A, Sampath V, Petroni D, Londei M, Nadeau KC. Phase 2a randomized, placebo-controlled study of anti-IL-33 in peanut allergy. JCI Insight. 2019 Nov 14;4(22):e131347. doi: 10.1172/jci.insight.131347. PMID 31723064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at two clinical sites in the United States between January, 2017 and March, 2018. Inclusion criteria included adult (older than 18 years) male or female participants with a clinical diagnosis of peanut allergy confirmed by an oral food challenge (OFC) at the screening visit (at 7-14 days before treatment).
Pre-assignment Details: On Day 1 eligible participants were randomized in a 3:1 ratio to receive one dose of either etokimab or placebo.
Groups:
- Etokimab: Participants received a single dose of 300 mg etokimab administered by 1-hour intravenous (IV) infusion on Day 1.
Period: Overall Study
Arm/Group | Etokimab | Placebo
Started | 15 | 5
Completed | 15 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomization Analysis Set included all randomized participants.
Groups:
- Etokimab: Participants received a single dose of 300 mg etokimab administered by 1-hour IV infusion on Day 1.
- Total: Total of all reporting groups
Arm/Group | Etokimab | Placebo | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (10.56) | 28.2 (13.14) | 30.0 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 4 | 13
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Cumulative Tolerated Peanut Dose During Oral Food Challenge [Mean (Standard Deviation); unit: mg] — Oral food challenges were performed at Baseline in accordance with the Practical Allergy (PRACTALL) consensus report. Escalating doses of peanut protein (peanut flour mixed with a non-allergic food vehicle such as apple sauce) consisting of 5, 20, 50, 100, 100, 100, and 125 mg (for a cumulative maximum dose of 500 mg) were given at 20 minute intervals. If the participant developed any signs of an objective allergic reaction, the challenge was stopped. The total cumulative tolerated dose of blinded peanut reached prior to reaction was recorded.
  mg | 250.3 (155.27) | 165.0 (151.66) | 229.0 (154.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. AEs include any clinical laboratory test results determined to be clinically significant by the investigator. AE was considered "serious" if there was any of the following outcomes: death, life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, other important medical events. Each AE was evaluated for severity (mild, moderate, or severe) and causal relationship to the study drug. AE was considered TEAE if the date of onset was during or after first dose of study treatment, or if the AE present at baseline worsened in either intensity or frequency after first dose of study treatment.
Time Frame: From first dose of study drug up to 45 days.
Population: Safety Analysis Set included all participants who received any portion of etokimab or placebo infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 15 | 5
Participants
  Any treatment-emergent adverse event (TEAE) | 15 | 5
  Serious TEAE | 0 | 0
  Mild TEAE | 3 | 0
  Moderate TEAE | 9 | 5
  Severe | 3 | 0
  TEAE related to study drug | 1 | 0
  Discontinued from the study due to TEAE | 0 | 0

2. Primary Outcome: Change From Baseline in Cumulative Tolerated Peanut Dose During Oral Food Challenge
Description: Oral food challenges were performed at Baseline and Day 14 in accordance with the Practical Allergy (PRACTALL) consensus report. Escalating doses of peanut protein (peanut flour mixed with a non-allergic food vehicle such as apple sauce) consisting of 5, 20, 50, 100, 100, 100, and 125 mg (for a cumulative maximum dose of 500 mg) were given at 20 minute intervals. If the participant developed any signs of an objective allergic reaction, the challenge was stopped. The total cumulative tolerated dose of blinded peanut reached prior to reaction was recorded.
Time Frame: Baseline and Day 14
Population: Full Analysis Set (FAS) included all participants who received etokimab or placebo who were present in the study until Day 14 with post-baseline OFC results.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 15 | 5
mg | 387.511 (39.053) | 327.466 (68.692)
Statistical Analysis 1: Comparison: Etokimab vs Placebo; Test type: Superiority; p = 0.463, ANCOVA; Analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline value as covariate; Least Squares (LS) Mean Difference = 60.046, 95% CI 2-sided [-108.566 to 228.657], Standard Error of Mean 79.918 — Treatment Difference = Etokimab - Placebo

3. Secondary Outcome: Change From Baseline in Oral Food Challenge Symptom Score at Day 14
Description: Oral food challenges were performed at Baseline and Day 14 in accordance with the PRACTALL consensus report.
  During OFC the OFC Symptom Scoring Assessment Tool was used to assess participants for common symptoms that can be suspected to be an allergic reaction involving the skin, upper respiratory, lower respiratory, gastrointestinal, and cardiovascular systems. Each symptom was scored according to the following scale: Grade 0 = sign or symptom not observed; Grade 1 = mild; Grade 2 = moderate, Grade 3 = severe. The score from each symptom was averaged to calculate the overall score at Baseline and on Day 14.
Time Frame: Baseline and Day 14
Population: FAS population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 15 | 5
score on a scale | 0.005 (0.008) | 0.004 (0.014)
Statistical Analysis 1: Comparison: Etokimab vs Placebo; Test type: Superiority; p = 0.962, ANCOVA; ANCOVA model with treatment as fixed effect and baseline value as covariate; LS Mean Difference = 0.001, 95% CI 2-sided [-0.031 to 0.032], Standard Error of Mean 0.016 — Treatment Difference = Etokimab - Placebo

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Etokimab
Description: The concentration of etokimab was measured using a validated assay method. The lower limit of quantification (LLOQ) was 0.400 microgram per milliliter (μg/mL).
Time Frame: Day 1 predose, 0.5 hours after the start of the infusion, end of infusion (EOI), 3 hours after EOI, 24, 96, 336 (Day 15), and 1056 (Day 45) hours after the start of infusion.
Population: Pharmacokinetic (PK) Analysis Set included all participants who received etokimab and had at least one post-dose serum concentration data value available for etokimab without any events or protocol deviation deemed to affect PK assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Etokimab
Number analyzed (Participants) | 15
μg/mL | 81.60 (22.9)

5. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Etokimab
Description: The concentration of etokimab was measured using a validated assay method. The lower limit of quantification (LLOQ) was 0.400 μg/mL.
Time Frame: Day 1 predose, 0.5 hours after the start of the infusion, EOI, 3 hours after EOI, 24, 96, 336 (Day 15), and 1056 (Day 45) hours after the start of infusion.
Population: PK Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | Etokimab
Number analyzed (Participants) | 15
hours | 1.080 [0.50 to 23.05]

6. Secondary Outcome: Area Under the Concentration-time Curve in Serum From Time Zero Extrapolated to Infinite Time (AUC0-inf) for Etokimab
Description: Area under the concentration-time curve in serum from time zero (predose) extrapolated to infinite time, calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration (Clast) divided by the apparent terminal rate constant (λz): AUC(0-last) + Clast/λz.
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (μg)*hour (h)/milliliter (mL)
Arm/Group | Etokimab
Number analyzed (Participants) | 15
microgram (μg)*hour (h)/milliliter (mL) | 15950 (27.8)

7. Secondary Outcome: Area Under the Concentration-time Curve in Serum From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) for Etokimb
Description: Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration, calculated by linear up/log down trapezoidal summation.
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Etokimab
Number analyzed (Participants) | 15
μg*h/mL | 14560 (25.6)

8. Secondary Outcome: Apparent Terminal Half-life (T1/2) for Etokimab
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Etokimab
Number analyzed (Participants) | 15
hours | 298.5 (18.3)

9. Secondary Outcome: Systemic Clearance for Etokimab
Description: Systemic clearance calculated as dose/ AUC(0-inf).
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Etokimab
Number analyzed (Participants) | 15
L/h | 0.01881 (27.9)

10. Secondary Outcome: Volume of Distribution at Steady State Following IV Dosing (Vss) for Etokimab
Description: Volume of distribution at steady state following intravenous dosing, calculated as mean residence time (extrapolated to infinity) multiplied by systemic clearance.
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Etokimab
Number analyzed (Participants) | 15
liters | 7.154 (19.8)

11. Secondary Outcome: Volume of Distribution (Vz)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Volume of distribution was estimated by dividing the systemic clearance by apparent terminal rate constant (λz).
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Etokimab
Number analyzed (Participants) | 15
liters | 8.096 (20.9)

12. Secondary Outcome: Apparent Terminal Rate Constant (λz)
Description: The terminal elimination rate constant (λz) is defined as the first-order rate constant describing the rate of decrease of drug concentration in the terminal phase. Apparent terminal rate constant was determined by linear regression of the terminal points of the log-linear concentration-time curve.
Time Frame: as for outcome 5
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Etokimab
Number analyzed (Participants) | 15
1/hour | 0.00231 (18.5)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 45
Arm/Group | Etokimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 15/15 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etokimab (N=15) | Placebo (N=5)
Hypersensitivity (Immune system disorders) | 14 | 5
Food allergy (Immune system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oral pruritus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Influenza like illness (General disorders) | 2 | 0
Adverse drug reaction (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Hangover (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02920021/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02920021/SAP_001.pdf